CLINICAL TRIAL: NCT05550428
Title: The Effects of Pulsed Electromagnetic Field Therapy on Patients With End-stage of Knee Osteoarthritis: A Double-blinded Randomized Control Trial
Brief Title: The Effects of Pulsed Electromagnetic Field Therapy on Patients With End-stage of Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022.185
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Sarcopenia
Keywords: Pulse electromagnetic field; PEMF; Knee Osteoarthritis; Knee OA; sarcopenia
MeSH Terms: conditions — Osteoarthritis, Knee; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into either treatment group or sham group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is doubled blinded, a subject 's specific ID card will be provided for each of the enrolled subject and the investigators don't know whether it is PEMF or Sham treatment for that subject's specific ID card. And the investigator will ask the manufactory about the number of grouping at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants in the intervention group will be exposed to PEMF treatment by a PEMF device (Quantum Tx, Singapore). Alternate legs will be exposed to PEMF treatment for 10 minutes per session, and the treatment regime will run biweekly for 8 weeks, summing up 16 sessions of PEMF exposure in total. All the participants were instructed on the proper performance of the exercise regimen by a senior physiotherapist before the commencement of the intervention. Subjects were then instructed to perform the home-based exercises on their own twice a week for eight weeks. One dedicated research assistant kept a weekly record of the participants' physical activity.
  Interventions: Other: home-based-exercise; Device: active pulsed electromagnetic field（PEMF）therapy
- Sham group (Sham Comparator): Participants in the intervention group will be exposed to PEMF treatment by a PEMF device (Quantum Tx, Singapore). Alternate legs will be exposed to PEMF treatment for 10 minutes per session, and the treatment regime will run biweekly for 8 weeks, summing up 16 sessions of sham exposure in total.All the participants were instructed on the proper performance of the exercise regimen by a senior physiotherapist before the commencement of the intervention. Subjects were then instructed to perform the home-based exercises on their own twice a week for eight weeks. One dedicated research assistant kept a weekly record of the participants' physical activity.
  Interventions: Other: home-based-exercise; Device: shame pulsed electromagnetic field（PEMF）therapy

INTERVENTIONS:
Other: home-based-exercise — All the participants were instructed on the proper performance of the exercise regimen by a senior physiotherapist before the commencement of the intervention. Subjects were then instructed to perform the home-based exercises on their own twice a week for eight weeks. One dedicated research assistant kept a weekly record of the participants' physical activity.
  sessions.
Device: active pulsed electromagnetic field（PEMF）therapy — Alternating legs on consecutive visits were exposed to either PEMF or sham therapy for eight weeks for a total of 16 PEMF sessions per participant, each leg receiving 8 exposures.
  Arms: Treatment group
Device: shame pulsed electromagnetic field（PEMF）therapy — Alternating legs on consecutive visits were exposed to either PEMF or sham therapy for eight weeks for a total of 16 sham PEMF sessions per participant, each leg receiving 8 exposures.
  Arms: Sham group

SUMMARY:
A double-blinded, randomizepd controlled trial to investigate the treatment effects of pulsed electromagnetic field (PEMF) on end stage of knee osteoarthritis patients with sarcopenia will be carried out. Subjects will be recruited from the Prince of Wales Hospital. Sixty participants age ≥ 60 will be invited to join this trial after informed consent. They will be randomised to any of the 2 groups: intervention group (n=30; PEMF (Quantum Tx) treatment), and control group (n=30; sham treatment with dummy exposure to PEMF). Both group will receive home-based exercise. Baseline measurements include appendicular muscle mass by DXA, bone microarchitecture (XtremeCT II), knee flexion and extension strength by handheld dynamometer, knee flexion and extension range of motion by goniometer, self-reported knee pain (VAS) and function by The Knee Injury and Osteoarthritis Outcome Score (KOOS), International Physical Activity Questionnaire (IPAQ) for assessment of physical activity level, quality of life by SF-36, hand grip test, bioelectrical impedance analysis （BIA）of body composition, postural stability, chair stand test, 30s arm curl test and 6-meter walking test. These measurements will be performed again at middle and end of treatment, 3, 6, and 12 months after commencement of treatment, except DXA, which will not be performed at the midpoint. In addition, blood samples will be taken at baseline, middle, and end of treatment, 3, 6, and 12 months after commencement of treatment, for determing of serum myokines which are reported to be sensitive to PEMF treatment and contribute to myogenesis.

The aim of this study is to conduct a double-blinded, randomized controlled trial to investigate the effects of PEMF treatment on muscle gain and pain relief in knee osteoarthritis with sarcopenia elderly in Hong Kong. We hypothesize that PEMF treatment is effective to promote a gain in muscle mass and function and pain relief in knee osteoarthritis with sarcopenia elderlies.

DETAILED DESCRIPTION:
PEMF therapy is the use of electromagnetic fields in a pulsating pattern directed towards the body.

The clinical use of PEMF therapies in orthopedics has been approved for over 40 years and commonly entail analgesic benefits. When specifically targeting the knee, however, evidence that the technology improves pain, physical function, and quality of life has been inconclusive, probably due to the unaddressed muscle weakness. Therefore, the approach employed in the present study was to target the leg musculature for its delivery of regenerative agents that naturally promote healing. The therapy entails a muscle-targeted, low-energy PEMF therapy previously used in human trials. Notably, this same PEMF paradigm was shown to improve functional mobility, increase lean muscle mass, and reduce pain in a community cohort containing frail elderly subjects. This PEMF paradigm has been demonstrated effective in promoting human muscle regeneration by inducing mitochondrial adaptations, similar to those invoked during oxidative muscle development in response to exercise

ELIGIBILITY:
Inclusion Criteria:

- subjects with knee osteoarthritis will be included:

1. radiographic Kellgren/Lawrence scale knee OA grade ≥3
2. enlistment on a TKR surgical waiting list; ability to comply with the trial assessments and fully comprehend questionnaires;
3. be over 50 years of age and
4. ability to walk unaided over 6 meters.

Exclusion Criteria:

* 1. With medical or musculoskeletal problems that could affect the ability to complete assessments (i.e. with walking aids or wheel-chaired).

  2. Severe cognitive impairments and neurological disorders that will affect data collection by questionnaires.

  3. Any medical conditions which are contraindicated to do exercise by PARQ restricting any physical activity.

  4. history of knee or hip surgeries 5. body mass index over 30 kg/m2 and 6. history of cancer.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
the change of knee extensor and flexor strength | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  The peak torque will be recorded in 2 trials in the 5 seconds isometric muscle strength test.

SECONDARY OUTCOMES:
the change of Muscle mass | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  Skeletal muscle mass will be measured by a Dual-energy X ray absorptiometry (DXA) scan or BIA according to standardized procedure The muscle mass in kg m^2 will be recorded in different time points.
the change of self-report knee pain and function | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  Self-reported pain and physical function will be measured using the the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire. This 42-item questionnaire is divided into five sub-scales, which address pain, other disease symptoms, function in activities of daily living, function in sport and recreation, and quality of life.
the change of 30s Arm curl | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  The participants receive a weight on the dominant hand. The weight is 2.27 kg [5 lb] for women and 3.63 kg [8 lb] for men. The task is to perform a 30s Arm Curl test. The number of the arm curl will be recorded.
the change of bone image | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  High-Resolution Peripheral Quantitative Computed Tomography Scans (HR-pQCT) High-resolution peripheral quantitative computed tomography scans (HR-pQCT) using XtremeCT II (Scanco Medical AG️, Brüttisellen, Switzerland) provides an analysis of bone microarchitecture at human peripheral sites with high spatial resolution and low exposure to radiation. Bone mineral density (BMD, calibrated with hydroxyapatite standards) and finite element analysis of subchondral bone over the knee joint will be performed using the Scanco software. Scans will be performed on both legs before the start of the PEMF treatment, in the middle of 8weeks, and after the completion of the PEMF treatment (3, 6- and 12-months).
the change of chair stand test | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  The rate of force development will be determined as the mean slope of the rising force of the first force peak of each of the 2nd to the 6th repetition in the interval of 30-70% exerted peak force. Results are reported as the mean of the two fastest approved trials in body weight per second (BW/s).
the change of postural stability | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  A force platform (Tekscan, U.S.) will be utilized to evaluate static postural control using the COP measures in static and dynamic postural control conditions. Sway path length (cm) of center of pressure (COP), velocity of COP (cm/s), ellipse area (cm^2)of COP (will be recorded.These static postural conditions include stand on double leg with open (DO) and close eyes (DC) for 30s, tandem stance for 30s, squat for 15s and stand on one leg with open eyes (SO) for 10s.Dynamic postural control will be evaluated using the task of transitioning from double-leg to single-leg standing.
the change of Serum myokine evaluation | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  Blood taking (5 ml) will be performed before PEMF treatment, and at 3, 6, and 12 months after the commencement of treatment. Serum will be prepared by centrifugation and kept in -80º freezer until use. Quantitative analysis for myokines and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme linked immunosorbent assay (ELISA). These include Brain-derived neurotrophic factor (BDNF), Fibroblast growth factor-21 (FGF-21), Interleukin-6 (IL-6), IL-15, Irisin, Myostatin (MSTN)/GDF8, Insulin-like growth factor 1 (IGF-1), FGF-2, IL-8, Follistatin, Musclin, Myonectin, Decorin, Meteorinlike, Osteopontin, Secreted protein acidic and rich in cysteine (SPARC), Klotho, Procollagen type III N-terminal peptide (P3NP), and C-terminal of troponin T1 (TNNT1)
the change of self-report pain | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  The Visual Analogue Scale (VAS) requires participants to rate participants' pain on a defined scale from 0-10 after each ending session of the PEMF therapy.
the change of self-report quality of life | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  Short Form-36 questionnaires (SF-36) will be used to evaluate Health-Related Quality of Life.
the change of physical activity | pre, mid, end of PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF]
  Physical Activity Readiness Questionnaire (PAR-Q) and International Physical Activity Questionnaire (IPAQ) will be used to determine whether participants should complete medical evaluation before participating in the exercise program in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun Ong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers

REFERENCES:
- [Derived] Wang QW, Ong MT, Man GC, Franco-Obregon A, Choi BC, Lui PP, Fong DTP, Qiu JH, He X, Ng JP, Yung PS. The effects of pulsed electromagnetic field therapy on muscle strength and pain in patients with end-stage knee osteoarthritis: a randomized controlled trial. Front Med (Lausanne). 2024 Oct 16;11:1435277. doi: 10.3389/fmed.2024.1435277. eCollection 2024. PMID 39478814